CLINICAL TRIAL: NCT06102226
Title: Deep Learning Algorithm for Detecting Obstructive Coronary Artery Disease Using Fundus Photographs
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yong Zeng (Other)
Responsible Party: Sponsor-Investigator, Yong Zeng, Beijing Anzhen Hospital, Beijing Anzhen Hospital
Organization: Beijing Anzhen Hospital (Other)
Other Study IDs: 121100004006885458
Record Dates: First submitted 2023-10-22; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Coronary Artery Disease; Artificial Heart Device User
MeSH Terms: conditions — Coronary Artery Disease | interventions — Coronary Angiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- coronary artery disease group / non- coronary artery disease group: Recruited patients were categorized into a coronary artery disease group and a non-coronary artery disease group on the basis of coronary angiography findings, and the presence of CAD was defined as the presence of a coronary artery lesion with a stenosis
  Interventions: Diagnostic Test: coronary artery imaging (coronary CTA or coronary angiography)

INTERVENTIONS:
Diagnostic Test: coronary artery imaging (coronary CTA or coronary angiography) — In order to obtain the gold standard labeling for coronary heart disease, this topic will form a panel of experts on labeling, and the diagnosis will be based on coronary angiography, defined as a lesion with a stenosis of at least 50% in at least one coronary artery

SUMMARY:
Artificial Intelligence, trained through model learning, can quickly perform medical image recognition and is widely used in early disease screening and assisted diagnosis. With the continuous optimization of deep learning, the application of AI has helped to discover some previously unknown associations with other systemic diseases. Artificial intelligence based on retinal fundus images can be used to detect anemia, hepatobiliary diseases, and chronic kidney disease, and to predict other systemic biomarkers. The above studies provide a theoretical basis for the application of artificial intelligence technology based on retinal fundus images to the diagnosis and prediction of cardiovascular diseases.

At present, there is still a lack of accurate, rapid, and easy-to-use diagnostic and therapeutic tools for predictive modeling of coronary heart disease risk and early screening tools in China and the world. Fundus image is gradually used as a tool for extensive screening of diseases due to its special connection with blood vessels throughout the body, as well as easy access, cheap and efficient. It is of great scientific and social significance to develop and validate a model for identification and prediction of coronary heart disease and its risk factors based on fundus images using AI deep learning algorithms, and to explore the value of AI fundus images in assisting coronary heart disease diagnosis and screening for a wide range of applications.

ELIGIBILITY:
Inclusion Criteria:

Eligible participants were ≥ 18 years of age, with clinically suspected CAD, and were scheduled for coronary angiography.

Exclusion Criteria:

The exclusion criteria were as follows: (i) prior percutaneous coronary intervention (PCI); (ii) prior coronary artery bypass graft (CABG); (iii) other heart disease (e.g., congenital heart disease, valvular heart disease, or macrovascular disease); (iv) inability to have photographs taken; and (v) and a diagnosis of ST-segment elevation myocardial infarction (STEMI). Prior to the coronary angiography procedure, all eligible patients provided informed consent to participate in the study and to have their photographs used for research purposes.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Eligible participants were ≥ 18 years of age, with clinically suspected CAD, and were scheduled for coronary angiography
Sampling Method: Probability Sample
Enrollment: 7000 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
AUC | December 30, 2024
  To evaluate the algorithm performance area under the receiver operating characteristic curve (AUC) were calculated

SECONDARY OUTCOMES:
sensitivity | December 30, 2024
  To evaluate the algorithm performance, the sensitivity were calculated
specificity | December 30, 2024
  To evaluate the algorithm performance, the specificity were calculated

CONTACTS AND LOCATIONS:
Overall Officials: Yong Zeng, Principal Investigator — Beijing An Zhen Hospital: Capital Medical University Affiliated Anzhen Hospital
Locations (1):
- Yong Zeng, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ye Y, Feng W, Ding Y, Chen Q, Zhang Y, Lin L, Xia P, Ma T, Ju L, Wang B, Chang X, Wang X, Cai L, Ge Z, Zeng Y. Retinal image-based deep learning for mild cognitive impairment detection in coronary artery disease population. Heart. 2025 Oct 14;111(21):1013-1019. doi: 10.1136/heartjnl-2024-325486. PMID 40379470